CLINICAL TRIAL: NCT00764140
Title: Insulin-like Growth Factors (IGF) Axis (IGFs, Its Binding Proteins,Receptors), Transforming Growth Factor Alpha and Beta 1 and Epidermal Growth Factor in the Urine and Serum of Patients With Hepatocellular Carcinoma.
Brief Title: Tumor Growth Factors in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Fa,Tsai, Professor of Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-960010
Record Dates: First submitted 2008-02-26; First posted 2008-10-01 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: tumor growth factor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and/or urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: Specific tumor growth factors (IGFs, its binding proteins,receptors; transforming growth factor alpha and beta 1 and epidermal growth factor) in the urine and serum will be measured in patients with hepatocellular carcinoma and healthy controls
- 1: Patients with hepatocellular carcinoma and Healthy controls
  Interventions: Biological: tumor growth factor concentration

INTERVENTIONS:
Biological: tumor growth factor concentration — spot urine or blood collection will be used to measure specific tumor growth factor
  Other Names: urine concentration of tumor growth factor; serum concentration of tumor growth factor
  Groups: 1

SUMMARY:
Malignant cells frequently produce many tumor growth factors to autocidal or endocrinal proliferate growth, metastasis,or angiogenesis about tumor cells. By studying tumor growth factors in hepatocellular carcinoma, one may know the tumor behavior, its relationship with clinical manifestation or invasion, and could be used as diagnostic or prognostic tools.This study aims to study the relationship between tumor growth factors in HCC ant its clinical relevance.

DETAILED DESCRIPTION:
The clinical relevance of patients will be evaluated by the concentrations of tumor growth factors.

ELIGIBILITY:
Inclusion Criteria:

* Histology proven HCC

Exclusion Criteria:

* No definitely diagnosed tumor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aspiration cytology or biopsy proved HCC and sex- and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
mortality | 5 years

SECONDARY OUTCOMES:
distant metastasis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Fa Tsai, M.D., Ph.D., Principal Investigator — Professor of Medine, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan